CLINICAL TRIAL: NCT01180309
Title: Lingual Frenum and Possible Alterations in the Articulation of Phonemes
Brief Title: Lingual Frenum and Articulation of Phonemes
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Collaborators: Izabella Santos Nogueira de Andrade (Unknown)
Responsible Party: REBEKA FERREIRA PEQUENO LEITE
Other Study IDs: RLeite
Record Dates: First submitted 2010-08-04; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Speech Disorders
Keywords: Tongue frenum; Lingual frenum; Audio Phonology; Speech disorders
MeSH Terms: conditions — Speech Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lingual frenum alterations: individuals each one with their phonological system complete

SUMMARY:
Purpose To investigate the relationship between lingual frenum and possible alterations in the articulation of phonemes.

Methods This is a quantitative observational study, the individual operative kind with transversal time reference. The population sample consisted of 16 individuals, each one with their phonological system complete. The data were captured through an application form that contained relevant aspects as to the qualitative-classification of the lingual frenum, quantitative-relation of mouth opening, with and without the tongue in the papillae, tongue mobility and ERT - 78 phonologically balanced words.

DETAILED DESCRIPTION:
The data were captured through an application form that contained relevant aspects as to the qualitative-classification of the lingual frenum, quantitative-relation of mouth opening, with and without the tongue in the papillae, tongue mobility and ERT - 78 phonologically balanced words.

ELIGIBILITY:
Inclusion Criteria:

* patients with the frenulum of the tongue - the presence of the central incisors and upper and lower side

Exclusion Criteria:

* patients in speech therapy aimed at enabling oral motor or speech - without integrity orofacial motor - patients using grid palate - with changes in the temporomandibular joint - anterior open bite

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The total study population consisted of subjects with complete phonological system, ie more than seven years of chronological age, both male and female, accompanied in the field of Dentistry, University of Fortaleza - UNIFOR.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Relation between lingual frenulum altered and articulation phonetics
  The quantitative assessment, we could classify the lingual frenulum as normal, values above 60%; questions to amend the frenulum-values between 50% and 60% and changed (short and / or anterior)-values below 50%.
  Finally, we carried out the assessment phonetics (AF) and it was applied Exam 12 Phonetic-Phonological ERT. This test, is composed of 78 pictures phonologically balanced, lexical repertoire familiar to the individual and easily recognizable pictorial.

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry, University of Fortaleza, Fortaleza, Ceará, Brazil